CLINICAL TRIAL: NCT06339060
Title: An Organ Preservation Strategies After Chemoradiotherapy Combined With Immunotherapy for Esophageal Cancer vs Cross Therapy.
Brief Title: An Organ Preservation Strategies After Chemoradiotherapy Combined With Immunotherapy for Esophageal Cancer (PALACE3).
Acronym: PALACE3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Prof, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTS-022
Record Dates: First submitted 2024-03-16; First posted 2024-04-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Cancer
Keywords: Chemoradiotherapy; Immunotherapy; Organ preservation; Active surveillance
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Masking Description: Randomize patients who meet the inclusion criteria Grouping, randomly assigned to the experimental group in a 1:1 ratio (organ preservation strategy after neoadjuvant chemotherapy combined with immunotherapy) And the control group (limited time for esophageal cancer radical surgery after neoadjuvant radiotherapy and chemotherapy)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1 Organ preservation (Experimental): A: Camrelizumab 200mg IV on days 1 and 22 B: Carboplatin (AUC=2) IV and Paclitaxel-albumin (50mg/m²) IV on day 1,8,15,22,29.
  C: Radiotherapy will start on day 1 of chemotherapy. A total of 41.4 Gy, 23 fractions of 1.8 Gy, 5 fractions a week.
  A+B+C=neoadjuvant therapy Patients will undergo clinical response evaluations (CREs) after neoadjuvant therapy(A+B+C）, If cancer is detected, surgery will be performed. Patients with clinical complete response （cCR） are eligible for active surveillance where regular CREs are performed to detect regrowth of cancer.Postoperative adjuvant therapy will follow the NCCN guideline.
  Interventions: Combination Product: Experimental: Arm 1 Organ preservation
- Arm 2 Surgery (Active Comparator): A: Camrelizumab 200mg IV on days 1 and 22 B: Carboplatin (AUC=2) IV and Paclitaxel-albumin (50mg/m²) IV on day 1,8,15,22,29.
  C: Radiotherapy will start on day 1 of chemotherapy. A total of 41.4 Gy, 23 fractions of 1.8 Gy, 5 fractions a week.
  Oesophagectomy will be offered to patients without contraindication.Postoperative adjuvant therapy will follow the NCCN guideline.
  Interventions: Combination Product: Active Comparator: Arm 2 Surgery

INTERVENTIONS:
Combination Product: Experimental: Arm 1 Organ preservation — Arm 1 patients will undergo clinical response evaluations (CREs) after neoadjuvant therapy(A+B+C）, If cancer is detected, surgery will be performed. Patients with clinical complete response （cCR） are eligible for active surveillance where regular CREs are performed to detect regrowth of cancer.Postoperative adjuvant therapy will follow the NCCN guideline.
  A: Camrelizumab 200mg IV on days 1 and 22 B: Carboplatin (AUC=2) IV and Paclitaxel-albumin (50mg/m²) IV on day 1,8,15,22,29.
  C: Radiotherapy will start on day 1 of chemotherapy. A total of 41.4 Gy, 23 fractions of 1.8 Gy, 5 fractions a week.
  A+B+C=Neoadjuvant therapy
  Arms: Arm1 Organ preservation
Combination Product: Active Comparator: Arm 2 Surgery — Arm 2 patients will undergo surgery after neoadjuvant therapy(B+C）.Postoperative adjuvant therapy will follow the NCCN guideline.
  B: Carboplatin (AUC=2) IV and Paclitaxel-albumin (50mg/m²) IV on day 1,8,15,22,29.
  C: Radiotherapy will start on day 1 of chemotherapy. A total of 41.4 Gy, 23 fractions of 1.8 Gy, 5 fractions a week.
  Arms: Arm 2 Surgery

SUMMARY:
Patients with locally advanced esophageal squamous cell carcinoma will randomly assigned to receive neoadjuvant chemo-radiotherapy combined with immunotherapy post organ preservation strategy (experimental group) or neoadjuvant chemo-radiotherapy followed by surgery (control group).

The 3-year overall survival rate is the primary outcome.

DETAILED DESCRIPTION:
The investigators will conduct the open, multicenter, prospective, randomized controlled clinical study(PALACE3). Patients with locally advanced esophageal squamous cell carcinoma will randomly assigned to either receive neoadjuvant synchronous radiotherapy and chemotherapy combined with immunotherapy followed by organ preservation strategy (experimental group, Arm1) or neoadjuvant concurrent radiotherapy and chemotherapy followed by radical surgery (control group,Arm 2). Collect relevant data on preoperative treatment, re examination after neoadjuvant therapy, perioperative and long-term follow-up of patients, and evaluate the clinical treatment effects (cCR rate), surgical pathological results (pCR rate, R0 resection rate, tumor regression grade, lymph node positivity rate), neoadjuvant therapy and perioperative complications, long-term oncological effects (total survival, disease-free survival), and quality of life of the two treatment plans through statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* A patient will be eligible for inclusion in this study only if ALL of the following criteria apply:

  * Histologically confirmed cT2-T4a,N0-N+,M0 resectable esophageal squamous cell carcinoma.
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-1
  * Patients approve and sign the informed consent

Exclusion Criteria:

* Patients with active autoimmune disease or history of autoimmune disease.
* Patients who have a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications.
* Subjects with a history of symptomatic interstitial lung disease.
* History of allergy to study drug components.
* Women must not be pregnant or breast-feeding.
* Men with female partners (WOCBP) that are not willing to use contraception.
* Patient has received prior chemotherapy, radiotherapy, target therapy and immune therapy for this malignancy or for any other past malignancy.
* medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival rate | From date of randomization until the date of death from any cause，up to 5 years
  The proportion of patients who survived within 3 years from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Hecheng Li, MD/PHD, Principal Investigator — Ruijin Hospital Shanghaijiaotong University School of Medicine
Locations (1):
- Ruijin hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided